CLINICAL TRIAL: NCT07267936
Title: Interventions for Maximizing Patient And Family Smoking Cessation Together
Acronym: IMPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P03172
Record Dates: First submitted 2025-05-22; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Smoking Cessation
Keywords: Household-based intervention; Smoking Cessation; Tobacco dependency
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: The intervention in this study involves inviting household members of the patients, to participate in the TTD program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with household members support (Experimental): Both the patients and the additional household members will be provided with Nicotine Replacement Therapy products and behavioural support. All participants will be followed up at 28 days, 3 months and 12 months post start Quit Date.
  The intervention in this study involves inviting household members of the patients, to participate in the Treating Tobacco Dependency program.
  The control group is patients without household members support. This is based on retrospective data of all patients who were admitted to Papworth Hospital and engaged with the Treating Tobacco Dependency Programme without any household members invited.
  Interventions: Other: Household member support

INTERVENTIONS:
Other: Household member support — The intervention in this study involves inviting household members of the patients, to participate in the Treating Tobacco Dependency program.

SUMMARY:
This feasibility study evaluates the effectiveness of a household-based smoking cessation intervention for patients and their household members. Patients who smoke and live with household members who also smoke will be invited to participate in the Treating Tobacco Dependency (TTD) program at Royal Papworth Hospital. The study aims to assess whether providing support to both patients and their household members improves quit rates and reduces relapse risk.

Participants will receive nicotine replacement therapy (NRT) and behavioural support, with follow-up assessments at 28 days, 3 months, and 12 months after starting the program. This study will compare outcomes to historical data from patients who participated in the TTD program without household support.

DETAILED DESCRIPTION:
The Treating Tobacco Dependency (TTD) program is currently available at Royal Papworth Hospital as part of an NHS initiative that started in August 2023. The program is available to all patients who smoke tobacco and are admitted to the hospital for at least 24 hours.

The TTD program provides NRT and behavioural counselling support, initially delivered by the TTD team at Royal Papworth Hospital, followed by HealthyYou, an NHS-approved stop smoking organization. Through this study, investigators are extending the invitation to household members of Royal Papworth Hospital patients to join the TTD program. This will allow the research team to assess whether a household-based intervention improves smoking cessation rates for both patients and their household members.

All participants will be followed up at 28 days, 3 months and 12 months post start of quit smoking. The smoking cessation rate will be compared to the routine TTD data set the research team has previously collected over the last year before household members were approached. This data will be acting as a control.

ELIGIBILITY:
Inclusion Criteria:

1. Any inpatient aged 18 and above admitted to Papworth Hospital who smoke. (Smoking is described as using any tobacco products as defined by the TTD programme)
2. Patient and household members must be eligible to join the TTD programme.
3. Patients must live in a household with other smokers.
4. Participants must live in Cambridgeshire and/or be registered with a GP Practice in the Cambridgeshire & Peterborough Integrated Care System

Exclusion Criteria:

1. Pregnant individuals - Pregnant individuals who smoke are offered a differing pathway to the standard TTD programme.
2. Contraindications for NRT.
3. Any household member who smokes unwilling to participate.
4. Individuals already enrolled on smoking cessation programme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Quit Rate among patients at 28 days | 28 days
  Assess difference in quit rates between patients with household support and the control group at 28 days.

SECONDARY OUTCOMES:
Patient relapse rate | 3 and 12 months
  Patient relapse rate at 3 and 12 months.
Household member quit rate | 28 days, 3 months and 12 months
  Household member quit rate at 28 days, 3 months and 12 months.
Difference in relapse rate between patients with and without household members support | 3 months and 12 months
  Difference in relapse rates between the two groups at 3 months and 12 months (Patients supported with household members and the control group)
Acceptance rate of support among household members | Baseline (At the time of screening , prior to enrollment)
  Potential household members who were approached but did not agree to participate in the study will be analyzed for the Acceptance of Support Among Household Members Who Smoke (%) endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Health Inequalities Specialist, Study Chair — Royal Papworth Hospital NHS Foundation Trust
Locations (1):
- Royal Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No